CLINICAL TRIAL: NCT06448273
Title: Phase I Clinical Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacokinetic Characteristics of Single and Multiple Doses of TQB3702 Tablets in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacokinetic of TQB3702 Tablets in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3702-I-02
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3702 tablets (Experimental): TQB3702 tables is administered as a single dose or multiple dose.
  Interventions: Drug: TQB3702 tablets
- TQB3702 placebo (Placebo Comparator): TQB3702 placebo is administered as a single dose or multiple dose.
  Interventions: Drug: TQB3702 placebo

INTERVENTIONS:
Drug: TQB3702 tablets — TQB3702 tablets is administered as a single dose on day 1, or once daily on Days 1 to 7 on multiple dose. Dosage: 100mg, 150/200mg.
  Arms: TQB3702 tablets
Drug: TQB3702 placebo — TQB3702 placebo contains no active substance.
  Arms: TQB3702 placebo

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled, dose-escalating clinical study aimed at evaluating the safety of TQB3702 tablets following single and multiple doses administered to healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants are aged between 18 and 55 years old (including 18 and 55 years old), regardless of gender;
* Male weight ≥50kg, female weight ≥45kg, with a body mass index (BMI) between 19 and 26 kg/m2;
* Fully understand this study, voluntarily participate in the trial, and have signed a written informed consent form;
* Subjects (including partners) are willing to self screen and voluntarily take appropriate and effective contraceptive measures (non contraceptive pills) within 6 months after the last study drug administration.

Exclusion Criteria:

* Pregnant and lactating women.
* Previous or current history of heart, endocrine, metabolic, kidney, liver, gastrointestinal, skin, infection, blood, neurological, or psychiatric diseases/abnormalities, or related chronic or acute diseases, the researcher assessed that it is not suitable to participate in the trial.
* Screening period vital signs, physical examination, laboratory examination, 15 lead electrocardiogram, chest anteroposterior lateral X-ray, abdominal ultrasound, female subjects also need to undergo uterine and bilateral accessory ultrasound, with abnormal and clinically significant results.
* There are serum virological abnormalities during the screening period;
* Active tuberculosis exists in the screening period, or is a close family contact of untreated active tuberculosis patients, or laboratory test T-SPOT.TB (a type of Enzyme-Linked Immunospot Assay) test positive individuals.
* Suffering from a history of severe bacterial, fungal, or viral infections within the first two months of randomization, requiring hospitalization and treatment with intravenous antibiotics or antiviral drugs.
* Randomly receive live vaccine within the first 4 weeks or plan to receive live vaccine during the study period.
* During the screening period, clinically significant infections may occur, including but not limited to upper respiratory tract infections, lower respiratory tract infections, urinary tract infections, etc., and require antibiotic or antiviral treatment.
* A history of severe herpes zoster or herpes simplex infection, including but not limited to herpes simplex encephalitis, disseminated herpes simplex, and generalized herpes zoster.
* Use any systemic cytotoxicity or systemic immunosuppressive drugs within the first 6 months of randomization or during the study period, or use any local cytotoxicity or local immunosuppressive drugs within the first 4 weeks of randomization or 5 half-lives or during the study period.
* Any other biological agents that have been marketed or studied within the first three months or five half-lives of randomization.
* Individuals who have undergone surgery within the first 4 weeks of randomization or plan to undergo surgery during the study period.
* Individuals who have lost blood or donated more than 400 mL of blood within the first 4 weeks of randomization.
* Individuals who have experienced external injuries within the first 6 months of randomization, such as car accidents, fractures, etc.
* Within the first 4 weeks of randomization, any prescription, over-the-counter, or herbal medication was taken, except for vitamin products.
* Potential difficulty in blood collection, with a history of fainting from needles and blood.
* Allergy to any known ingredients of TQB3702, or any history of severe drug allergies.
* Individuals with a history of drug abuse or positive urine drug screening.
* Smoking more than 5 cigarettes per day or using an equivalent amount of nicotine or nicotine containing products within the first 3 months of randomization, or not stopping the use of any tobacco products during the trial period.
* Individuals who have long-term alcohol abuse or have consumed more than 14 units of alcohol per week within the first 3 months of screening, or have been unable to abstain from alcohol during the trial period, or have tested positive for alcohol breath.
* Any other reasonable medical, mental, or social reasons that the researcher believes cannot participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events rate | 17 days
  Number of subjects with adverse events (AEs) and serious adverse events (SAEs), the evaluation criteria for the nature and severity of adverse events are based on the National Cancer Institute's CommonTerminology Criteria for Adverse Events (NCI CTCAE version 5.0).
Abnormal laboratory test indicators | 17 days
  Number of subjects with clinically significant abnormalities in vital signs, electrocardiogram (ECG), and laboratory parameters graded by CTCAE v5.0.

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (Tmax) | 1 hour (pre-dose), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 1 for sing dose and multiple dose. 0.5 hour pre-dose of day 4 to day 7, and 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 7 for multiple dose
  Time to reach maximum (peak) plasma concentration following drug administration.
Maximum Plasma Concentration (Cmax) | 1 hour (pre-dose), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 1 for sing dose and multiple dose. 0.5 hour pre-dose of day 4 to day 7, and 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 7 for multiple dose
  The Cmax is the maximum observed plasma concentration of TQB3702.
Elimination half-life (t1/2) | 1 hour (pre-dose), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 1 for sing dose and multiple dose. 0.5 hour pre-dose of day 4 to day 7, and 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours post-dose of Day 7 for multiple dose
  Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China